CLINICAL TRIAL: NCT05471401
Title: GI Organ Tracking Via Balloon Applicators
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202207133
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer; Kidney Cancer; Larynx Cancer; Liver Cancer; Lung Cancer; Digestive Organs--Cancer; Intrathoracic--Cancer; Respiratory Organs--Cancer; Pancreas Cancer; Small Intestine Cancer; Stomach Cancer; Colon Cancer; Rectal Cancer
Keywords: Gastric balloon
MeSH Terms: conditions — Esophageal Neoplasms; Kidney Neoplasms; Laryngeal Neoplasms; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Occlusion balloon catheter (Experimental): -Each participant will have an embolectomy balloon that is FDA approved for peripheral and neurovasculature temporary occlusion placed by nose or mouth. Anatomical position of balloon will be verified by on-board MR or CT imaging in to assess feasibility of using a duodenal balloon in this population. Participants who are imaged on the MR treatment machine will also be imaged with 4 or 8 frame per second sagittal imaging to assess real-time stomach and balloon respiratory motion. Participants imaged on CT based imaging (i.e. Ethos/Halcyon ring gantry system) will have CBCTs acquired at timed intervals (approximately 5-10 minutes between scans). After imaging, the balloon will be deflated and removed at that time.
  Interventions: Device: Balloon-tipped catheter

INTERVENTIONS:
Device: Balloon-tipped catheter — Gastric balloon

SUMMARY:
The hypothesis of this study is that an occlusion balloon catheter placed in the stomach via an oral or nasogastric route will be safe and permit tracking of the stomach during radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive intra-thoracic or abdominal radiation therapy. It is not required that the stomach be in the radiation field.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior trauma or surgical intervention that would alter the anatomy of the upper airs (nasogastric route), esophagus or stomach.
* Previous complete or partial surgical resection of the esophagus, stomach, or duodenum.
* Presence of implantable devices (e.g., automatic internal cardiac defibrillator, cardiac or gastric pacemaker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who undergo successful inflation of the gastric balloon with oral contrast agent, with verification by MR or CT imaging | Completion of follow-up for all participants (estimated to be 1 year)

SECONDARY OUTCOMES:
Number of grade grade ≥ 2 adverse events that are probably or definitely associated with the balloon inflation | Completion of follow-up (estimated to be 4 weeks)
Translation movement of stomach between CBCT scans with and without balloon insufflation | Day of procedure (Day 1)
  -Stomach position will be compared between interval scans.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon review and approval of request by the upper-GI focus group leaders at Siteman Cancer Center.
Supporting Information: Study Protocol, SAP
Time Frame: Contact investigator for details.
Access Criteria: Contact investigator for details.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu